CLINICAL TRIAL: NCT05019586
Title: Helicobacter Pylori Resistance. A Study of Morbidity, Immunological and Clinical Phenotypes
Brief Title: Helicobacter Pylori Resistance
Acronym: CRIHEP
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Jon Florholmen, professor, MD, University Hospital of North Norway
Other Study IDs: University Hosp North Norway
Record Dates: First submitted 2021-08-14; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Helicobacter Pylori Resistance
Keywords: Gastrointestinal Symptom Rating Scale, Helicobacter pylori resistance, levofloxacin, Sydney score
MeSH Terms: interventions — Levofloxacin; Amoxicillin; Clarithromycin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — RNA measure of mucosal transcripts, mucosal histology, cultures including antibiotic sensitivity to HP from mucosal biopsies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Helicobacter pylori resistance: Patients with treatment resistance to Helicobacter pylori treatment registered at GI-unites from 1990-2012 and included from 2010 to 2012. These patients were treated with a triple therapy of levofloxacin, amoxicillin and proton inhibitor for 10 days
  Interventions: Drug: levofloxacin, amoxicillin, clarithromycin
- Newly diagnosed Helicobacter pylori: Patients with newly diagnosed Helicobacter pylori infection from 2010-2012.These patients were treated with a triple therapy of clarithromycin, amoxicillin and proton inhibitor for 10 days
  Interventions: Drug: levofloxacin, amoxicillin, clarithromycin
- Previously eradicated Helicobacter pylori infection: Patients with previously Helicobacter pylori infection included from 2010-2012.
- Never Helicobacter pylori infection: Patients with previously Helicobacter pylori infection included from 2010-2012.

INTERVENTIONS:
Drug: levofloxacin, amoxicillin, clarithromycin — Triple therapy of Helicobacter pylori including two antibiotics and a proton inhibitor for 10 days
  Groups: Helicobacter pylori resistance; Newly diagnosed Helicobacter pylori

SUMMARY:
The main goal of the study was to characterize the morbidity, immunological, microbiolical and clinical phenotypes of patients with treated- resistance to Helicobacter pylori (HP) infection, and the effect of triple therapy including the levofloxacin. Control groups were newly diagnosed, previously infected and never infected HP patients

DETAILED DESCRIPTION:
See Nestegard O, et al. PLOS ONE | https://doi.org/10.1371/journal.pone.0238944 September 23, 2020

ELIGIBILITY:
Inclusion Criteria:

Patients referred to a GI- unite with upper GI complains and performing an upper endoscopy -

Exclusion Criteria:

Patients with severe chronic diseases and not willing to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients referred to Gastrointestinal (GI) unite in the time periode from 1990 to 2010 and defined as resistant to triple Helicobacter pylori (HP) treatment
  2. Patients referred to GI unite in the time periode from 2010 to 2012 due to opper GI complaints. Included were patients a) newly diagnosed HP, b) previously successful triple HP therapy, and c) never HP infected
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2010-04-15 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Characterization of patients with chronic HP infection resistant to previous conventional triple therapy | 2010-2012
  Clinical data including endoscopy, histology, microbiological data including resistance measurements, immunological data (mucosal tranacrips), effect of triple therapy
Endoscopy | 2010-2012
  endoscopic description of mucosa bye endoscopy
Histology | 2010-2012
  Histological characterizations of inflammation (Sydney) of gastric mucosa
Immunology | 2010-2012
  Immunological mucosal characterizations of pro- and antiinflammatory cytokine transcript (PCR)
HP microbiology | 2010-2012
  HP microbiology sensitivity to metronidazol, amoxicillin, clarithromycine, levofloxacin and tetracycline

CONTACTS AND LOCATIONS:
Overall Officials: Jon Florholmen, Principal Investigator — Department of Gastroenterology, Norwegian Artic University/Universiuty of Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nestegard O, Moayeri B, Halvorsen FA, Tonnesen T, Sorbye SW, Paulssen E, Johnsen KM, Goll R, Florholmen JR, Melby KK. Helicobacter pylori resistance to antibiotics before and after treatment: Incidence of eradication failure. PLoS One. 2022 Apr 20;17(4):e0265322. doi: 10.1371/journal.pone.0265322. eCollection 2022. PMID 35442962